CLINICAL TRIAL: NCT07269405
Title: A Randomised Controlled Trial of a Multi-component Postpartum Intervention to Prevent Dysglycemia in Women With a History of Gestational Diabetes Mellitus (GDM)
Brief Title: Study to Prevent Dysglycemia in Women With GDM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Ronald C.W. Ma, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2025.127
Record Dates: First submitted 2025-10-02; First posted 2025-12-08 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Gestatiaonl Diabetes Mellitus; GDM
Keywords: Gestatiaonl diabetes mellitus; GDM; Postpartum; Lifestyle intervention
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: Multi-component lifestyle intervention
Who Masked: Investigator, Outcomes Assessor
Masking Description: Data analysts
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Lifestyle Intervention (Experimental): Multicomponent intervention include e-care and wearables
  Interventions: Behavioral: Intervention
- Conventional Care (Other): Conventional care
  Interventions: Other: Conventional care

INTERVENTIONS:
Behavioral: Intervention — The intervention groups will receive information on basic dietary information and have access to e-platform.
  Participants will attend individualised/ group dietary counselling sessions biweekly in the first 4 months during the intensive phase and thereafter bimonthly and biyearly between year 1 to year 3.
  This will include 16 sessions with a dietitian/nutritionist and 4 sessions with an exercise instructor. Participants will be given an individualized menu plan aiming at achieving a varied balanced diet with an emphasis on fibre intake and moderate-carbohydrate, low-fat, low-glycaemic index products in appropriate portions.
  Arms: Multicomponent Lifestyle Intervention
Other: Conventional care — The control group will receive basic dietary information leaflets and will have access to the e-care platform for the three-year period. The control group will receive routine lifestyle advice.
  Arms: Conventional Care

SUMMARY:
Women with a history of gestational diabetes mellitus (GDM) have a 7-fold increased risk of type 2 diabetes (T2D), with the risk at its highest during the 3-6 years postpartum. GDM thus represents one of the strongest known risk factors for T2D.

Only 30-60% of women with GDM returned for postpartum visits, with the majority defaulting on postpartum glucose tolerance testing. Women with GDM also have an increased risk of hypertension, cardiovascular disease (CVD), non-alcoholic fatty liver disease, and other comorbidities. Through this study, participants will receive lifestyle advice that may help them prevent diabetes. The study will help determine whether a multicomponent intervention will prevent incident dysglycemia and improve offspring cardiometabolic health. This will inform healthcare professionals and policymakers if these interventions are helpful. The control group will receive basic dietary information leaflets and will have access to the e-care platform for the three-year period (8-166 weeks postnatal). They will receive routine lifestyle advice and counseling. The intervention groups will receive information on basic dietary information and have access to the e-platform. Participants will attend individualized/group dietary counseling sessions biweekly in the first 4 months during the intensive phase (V1-V7) and thereafter bimonthly (V8-10, 28-50 weeks postnatal) and biyearly between year 1 to year 3. This will include 16 sessions with a dietitian/nutritionist and 4 sessions with an exercise instructor. Participants will be given an individualized menu plan aiming at achieving a varied, balanced diet with an emphasis on fiber intake and moderate-carbohydrate, low-fat, low-glycemic index products in appropriate portions. The lifestyle intervention program will incorporate motivational interviewing and behavioral modification to enhance health knowledge on daily diet and physical activity. The lifestyle intervention aims to achieve targets on body weight, dietary intake, and physical activities.

DETAILED DESCRIPTION:
The high-risk nature of women with GDM highlights this group as the "low-hanging fruit" who would substantially benefit from engagement in diabetes prevention programs. Lifestyle intervention has been shown to reduce the progression to T2D among women with GDM.

In a systematic review and meta-analysis including 8 lifestyle intervention trials implemented post-GDM, there was a homogenous 25% reduction (relative risk (RR): 0.75; 95% confidence interval (CI) 0.55-1.03) in incident diabetes, though not statistically significant. Of note, trials offering intervention soon after delivery (i.e., <6 months postpartum) were most effective. This contrasts with efforts during pregnancy to reduce GDM, which have failed to reduce GDM unless initiated very early. The long-term follow-up of mothers and offspring from the Hyperglycemia and Adverse Pregnancy Outcome (HAPO) study has highlighted the increased risk of adiposity, obesity, and diabetes in offspring, who are at increased risk of NCDs later in life. Hence, enrolling mothers with GDM in empowerment and prevention programs will not only reduce their risk of diabetes and CVD but may also benefit other family members, in particular the offspring.

In a previous pilot lifestyle intervention trial in mothers with GDM in the postpartum setting (NCT03669887), the investigators established the logistics of engaging mothers during the busy postpartum period, performing repeated OGTTs and clinical assessments, and co-designing with mothers a lifestyle intervention curriculum suitable for implementation during the postpartum period. The investigators demonstrated the benefit of the intervention in improving the health behaviors of GDM mothers at 1 year. The investigators were able to engage participants with GDM and noted their misconceptions about the long-term impact of GDM, their concerns about whether they can breastfeed, and lack of awareness of the risk of obesity in their offspring. The intervention arm had improved dietary quality as measured using the Dietary Quality Index-International (DQI-I) score, more favorable changes in BMI at 6 months postpartum, and a trend towards better glycemic status after 12 months.

Objectives:

Primary objective

- To evaluate the effect of a multicomponent postpartum intervention to prevent incident dysglycemia in women with a history of GDM.

Secondary objectives"

* To evaluate the effect of a multicomponent intervention on body weight and composition.
* To evaluate the effect of a multicomponent intervention on cardiometabolic health parameters including blood pressure, heart rate, vital signs, and lipid profiles.
* To evaluate the effect of a multicomponent intervention on continuous glucose monitoring metrics.
* To evaluate the effect of a multicomponent intervention on dietary intake.
* To evaluate the effect of a multicomponent intervention on physical activity.
* To evaluate the effect of a multicomponent intervention on breastfeeding and infant feeding practices.
* To evaluate the effect of a multicomponent intervention on offspring growth, weight, and adiposity.

Compared with conventional care.

Study design: Multi-center, prospective, parallel-group, open-label randomized controlled trial Study population: Women with a history of GDM Sample size: 800 subjects Intervention: Multicomponent intervention including e-care and wearables Comparator: Conventional care

Setting:

Women with a history of gestational diabetes will be identified from antenatal clinics. The study will be conducted at the Prince of Wales Hospital and the CUHK Medical Centre.

ELIGIBILITY:
Inclusion Criteria:

1. Women with a history of gestational diabetes mellitus and one additional risk factor (obesity, family history of diabetes, impaired fasting glycemia and/or impaired glucose tolerance and/ and or risk understanding by yourself RUBY score of ≥ 8) at 6-12 weeks postpartum
2. Singleton pregnancy
3. Willingness, ability and commitment to comply with study procedures
4. In the opinion of the investigator, absence of any physical limitations, addictive diseases, or underlying medical conditions (including mental health) that may preclude the patient from being a suitable study candidate.
5. Normally residing in Hong Kong
6. Able to communicate in Chinese
7. Written informed consent to participate in the study provided by the patient

Exclusion Criteria:

1. Known current diabetes
2. Current or previous use of glucose-lowering or weight loss drugs at screening
3. Concurrent participation in other weight loss or lifestyle intervention programmes
4. Any active acute or chronic disease or condition that, in the opinion of the investigator, might interfere with the performance of this study
5. Any active acute or chronic infectious disease that, in the opinion of the investigator, would pose an excessive risk to study staff
6. Current use or recent exposure to any medication that in the opinion of the investigator could have an influence on the patient's ability to participate in this study or on the performance of the test device
7. Known uncontrolled thyrotoxicosis
8. Current use of steroids
9. Known current or recent alcohol or drug abuse
10. Currently participating in another investigational study protocol where the testing or results may interfere with study compliance, diagnostic results, or data collection
11. An identified protected vulnerable patient (including but not limited to those in detention, or a prisoner)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Proportion with deterioration in glycaemic status (ie. from NGT to pre-diabetes (IFG or IGT), or pre-diabetes to T2D, based on annual OGTT | 1 Year, 2 Year, 3 Year

SECONDARY OUTCOMES:
Fasting glucose and post challenge glucose | 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in fasting glucose and post challenge glucose
Body weight | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in body weight
BMI | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in BMI
Body composition | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in body composition
Systolic and diastolic blood pressure | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in systolic and diastolic blood pressure
Heart rate | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in heart rate
CGM metrics | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in CGM metrics, including times in range (TIR), above range, and below range
Physical activity levels (IPAQ) | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in physical activity levels assessed by IPAQ
Diet composition and quality (The FIGO Nutrition Checklist) | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in diet composition and quality assessed by The FIGO Nutrition Checklist
Lipid profiles | 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in lipid profiles
Proportion breastfed | End of intensive intervention period (Postnatal week 20-26) and 1 Year, 2 Year, 3 Year
  Difference between intervention and control groups in proportion of breastfed
Offspring weight | Postnatal week 160-166
  Difference between intervention and control groups in offspring weight
Offspring adiposity (skinfold thickness) | Postnatal week 160-166
  Difference between intervention and control groups in offspring adiposity (skinfold thickness)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Therapeutics, The Chinese University of Hong Kong (CUHK), Ward 3M, Diabetes and Endocrine Research Centre, 3/F Day Treatment Block and Children Wards (Old Block), Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
to further seek approval among project team